CLINICAL TRIAL: NCT06226389
Title: 2-Year Clinical Evaluation of Different Bulk-fill Resin Composite Restorative Systems in Posterior Teeth
Brief Title: Clinical Evaluation of Different Bulk-fill Composite Restorations on Posterior Teeth
Acronym: 2-Year
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A02011023
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-12

CONDITIONS: Carious Teeth
Keywords: Bulk-fill composite, posterior cavities
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 Different bulk-fill composite (Experimental): Bulk-fill composite will be applied in different 4 posterior cavities with 3-4 ml in depth
  Interventions: Procedure: 4 different bulk-fill composite
- Aging (Experimental): For long term follow up
  Interventions: Procedure: 4 different bulk-fill composite

INTERVENTIONS:
Procedure: 4 different bulk-fill composite — Posterior cavities either class 1/2

SUMMARY:
Different bulk-fill composites will be applied in different posterior cavities then compared

DETAILED DESCRIPTION:
Patients must be in middle age(25-55) age,able to regularly follow up,not pregnant and at least have 4 carious molars

ELIGIBILITY:
Inclusion Criteria:

* at least 4 carious molars

Exclusion Criteria:

* pregnancy patient
* Not able to regularly follow up
* bad oral hygiene

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-01-17 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Difference between baseline and after 2 years of evaluation of resin based composite | Baseline to 2 years
  Change in FDI criteria

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa S Elsaeed, Assistant lecturer, Principal Investigator — Assistant lecturer
Locations (1):
- Mansoura,Faculty of Dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Yes Study Protocol, Statistical Analysis Plan can be shared to other researchers
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after 2 years
Access Criteria: For anyone